CLINICAL TRIAL: NCT05772442
Title: Investigating the Metabolomic Profile of Transplanted Heart With and Without Pathological Signs of Rejection
Brief Title: Cardiac Transplant Metabolomics With and Without Rejection
Acronym: ANTIPARTICLE
Status: Not yet recruiting | Type: Observational
Sponsor: Western University, Canada (Other)
Collaborators: Canadian Cardiovascular Society (Other); Bayer (Industry); University of Alberta (Other); Queen's University (Other)
Responsible Party: Sponsor
Other Study IDs: 122451
Record Dates: First submitted 2023-03-05; First posted 2023-03-16 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Heart Transplant Rejection
Keywords: Transplant; Metabolomics; Rejection
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No pathological signs of rejection: Routine endomyocardial biopsy did no show pathological signs of rejection (0R) based on the International Society for Heart and Lung Transplantation (ISHLT) 2004 acute cellular rejection grading scheme.
  Interventions: Diagnostic Test: Extra blood samples (5-10 mL) drawn
- With pathological signs of rejection: Routine endomyocardial biopsy showed pathological signs of rejection (1R, 2R, and 3R) based on the International Society for Heart and Lung Transplantation (ISHLT) 2004 acute cellular rejection grading scheme.
  Interventions: Diagnostic Test: Extra blood samples (5-10 mL) drawn

INTERVENTIONS:
Diagnostic Test: Extra blood samples (5-10 mL) drawn — Extra blood samples will be sent for metabolomics analysis.

SUMMARY:
Patient who received a heart transplant may develop organ rejection. Currently, an invasive biopsy of the heart needs to be performed to diagnose rejection. The purpose of this research study is to identify novel metabolic biomarkers that can be developed into a blood test that can identify signs of rejection without doing a heart biopsy.

DETAILED DESCRIPTION:
Background:

Cardiac transplantation remains the treatment of choice for end-stage heart failure. Rejection is a major risk factor affecting the outcome and survival in transplant recipients. Endomyocardial biopsy is the gold standard for diagnosis of post-transplantation rejection, but it is an invasive procedure with potential serious complications. Moreover, due to limited catheterization lab time and time required to process biopsied tissue, the transplanted organs could potentially receive irreversible damages upon diagnosis of acute rejection. Current available non-invasive test involving detecting donor DNA in recipient's blood is still costly and has many limitations. Hence, a better non-invasive and timely diagnostic approach with high sensitivity and specificity is needed to help improve the diagnosis of acute post-cardiac transplant rejection.

Methods At the London Health Science Centre, patient who had a cardiac transplant will undergo routine weekly blood sample collection and endomyocardial biopsy for the first 4 weeks to screen for acute rejection. After informed consent was obtained for routine endomyocardial biopsy and research study, endomyocardial tissue samples and blood will be collected from the patient. Two to three biopsy samples and the blood were processed according to the protocols provided by the Metabolomic Innovation Centre (Edmonton, Alberta, Canada). The sample will be analyzed using the high-performance chemical isotope labelling liquid chromatography mass spectrometry metabolomics platform.

Expected Results:

Using the non-targeted metabolomics, the primary objective is to identify promising novel candidate biomarkers from the blood samples that can help us identify patients who are in acute rejection post-cardiac transplant. The blood sample biomarkers can be validated with endomyocardial biopsy metabolomics data. In addition, characterizing the metabolic profile of transplanted heart can provide insights for the myocardial energetics in transplanted heart. These data can potentially help physicians predict the likelihood of patients developing rejection.

Conclusion:

Metabolomics is an emerging technology used for absolute quantification of metabolites in tissues, cells, and biological fluids based on mass spectrometry. Investigators are hoping to use this technology to identify novel candidate biomarkers that can be used to accurately predict the presence of acute rejection in post-cardiac transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients with heart transplant undergoing routine endomyocardial biopsy and blood work for transplant rejection screening and workup.
* Patients or substitute decision makers are able to provide informed consent to agree to participate in this study.

Exclusion Criteria:

* Patients or substitute decision makers declined to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had cardiac transplant undergoing routine blood work and endomyocardial biopsy in the catheterization lab at London Health Sciences Centre - University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Metabolomics differences detected in the blood sample of patient with signs of transplant rejection vs. no rejection. | 1-2 year to obtain these samples.
  25 blood samples in the no rejection group and 25 blood samples in the rejection group will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Smith, MD, Principal Investigator — Western University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andrew J, Macdonald P. Latest developments in heart transplantation: a review. Clin Ther. 2015 Oct 1;37(10):2234-41. doi: 10.1016/j.clinthera.2015.08.019. PMID 26497799
- [Background] Almenar L, Cardo ML, Martinez-Dolz L, Garcia-Palomar C, Rueda J, Zorio E, Arnau MA, Osa A, Palencia M. Risk factors affecting survival in heart transplant patients. Transplant Proc. 2005 Nov;37(9):4011-3. doi: 10.1016/j.transproceed.2005.09.160. PMID 16386612
- [Background] Cooper LT, Baughman KL, Feldman AM, Frustaci A, Jessup M, Kuhl U, Levine GN, Narula J, Starling RC, Towbin J, Virmani R; American Heart Association; American College of Cardiology; European Society of Cardiology; Heart Failure Society of America; Heart Failure Association of the European Society of Cardiology. The role of endomyocardial biopsy in the management of cardiovascular disease: a scientific statement from the American Heart Association, the American College of Cardiology, and the European Society of Cardiology. Endorsed by the Heart Failure Society of America and the Heart Failure Association of the European Society of Cardiology. J Am Coll Cardiol. 2007 Nov 6;50(19):1914-31. doi: 10.1016/j.jacc.2007.09.008. No abstract available. PMID 17980265
- [Background] Zwang NA, Turka LA. Transplantation immunology in 2013: New approaches to diagnosis of rejection. Nat Rev Nephrol. 2014 Feb;10(2):72-4. doi: 10.1038/nrneph.2013.262. Epub 2013 Dec 17. PMID 24342957
- [Background] CHIBA C, WOLF PL, GUDBJARNASON S, CHRYSOHOU A, RAMOS H, PEARSON B, BING RJ. Studies on the transplanted heart. Its metabolism and histology. J Exp Med. 1962 Apr 1;115(4):853-66. doi: 10.1084/jem.115.4.853. PMID 13878918
- [Background] Kolwicz SC Jr, Purohit S, Tian R. Cardiac metabolism and its interactions with contraction, growth, and survival of cardiomyocytes. Circ Res. 2013 Aug 16;113(5):603-16. doi: 10.1161/CIRCRESAHA.113.302095. PMID 23948585
- [Background] Akki A, Smith K, Seymour AM. Compensated cardiac hypertrophy is characterised by a decline in palmitate oxidation. Mol Cell Biochem. 2008 Apr;311(1-2):215-24. doi: 10.1007/s11010-008-9711-y. Epub 2008 Feb 16. PMID 18278440
- [Result] Lin F, Ou Y, Huang CZ, Lin SZ, Ye YB. Metabolomics identifies metabolite biomarkers associated with acute rejection after heart transplantation in rats. Sci Rep. 2017 Nov 13;7(1):15422. doi: 10.1038/s41598-017-15761-3. PMID 29133921
- [Result] Xiong PY, Motamed M, Chen KH, Dasgupta A, Potus F, Tian L, Martin A, Mewburn J, Jones O, Thebaud A, Archer SL. Inhibiting pyruvate kinase muscle isoform 2 regresses group 2 pulmonary hypertension induced by supra-coronary aortic banding. Acta Physiol (Oxf). 2022 Feb;234(2):e13764. doi: 10.1111/apha.13764. Epub 2022 Jan 17. PMID 34978755
- [Result] Xiong PY, Tian L, Dunham-Snary KJ, Chen KH, Mewburn JD, Neuber-Hess M, Martin A, Dasgupta A, Potus F, Archer SL. Biventricular Increases in Mitochondrial Fission Mediator (MiD51) and Proglycolytic Pyruvate Kinase (PKM2) Isoform in Experimental Group 2 Pulmonary Hypertension-Novel Mitochondrial Abnormalities. Front Cardiovasc Med. 2019 Jan 25;5:195. doi: 10.3389/fcvm.2018.00195. eCollection 2018. PMID 30740395